CLINICAL TRIAL: NCT06353685
Title: A Phase II Clinical Study of Continuous Hyperfractionated Accelerated Radiotherapy(CHART) in Oral Cancer Patients Who Underwent Neoadjuvant Chemotherapy Combined With Immunotherapy and Achieved pCR and MPR After Surgery.
Brief Title: De-Escalation Postoperative Radiotherapy for Oral Squamous Cell Carcinoma With pCR/MPR.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhuofei Bi, Associate Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-238-01
Record Dates: First submitted 2024-03-23; First posted 2024-04-09 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: De-escalated Radiotherapy; Head and Neck Cancer
Keywords: de-escalated radiotherapy; CHART; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous hyperfractionated accelerated radiotherapy(CHART) (Experimental)
  Interventions: Radiation: Continuous, hyperfractionated, accelerated radiotherapy(CHART)

INTERVENTIONS:
Radiation: Continuous, hyperfractionated, accelerated radiotherapy(CHART) — high-risk CTV area (CTV1), 45Gy in total, fraction dose of 1.5Gy, twice a day, bioequivalent dose (BED) of 51.75Gy; Low-risk CTV area(CTV2), 39Gy in total , fraction dose of 1.3Gy, twice a day, BED of 44.07Gy; A total of 30 radiotherapy fraction were performed 10 times a week for 3 weeks.

SUMMARY:
The prognosis of locally advanced oral squamous cell carcinoma(OSCC ) is poor, and there are still many problems to be solved in the current treatment paradigm. Neoadjuvant chemotherapy combined with immunotherapy can significantly improve the pCR and MPR rates in patients with locally advanced OSCC. For patients who achieve pCR and MPR after neoadjuvant therapy and surgery, it is still hotly debated regarding whether to implement postoperative de-escalation radiotherapy. Neoadjuvant therapy is an ideal predictor of radiosensitivity. In theory, neoadjuvant therapy can eliminate microscopic lesions, thereby reducing the dose and volume of irradiation.

Continuous hyperfractionated accelerated radiotherapy (CHART, based on hyperfractionated radiotherapy, increasing daily or weekly treatments and shortening the total treatment duration, but reducing the total dose), is to give a higher dose of radiation to tumor tissue in a shorter period of time, so as to overcome the accelerated reproliferation and inhibit the repair of sublethal damage of tumor cells. It is beneficial to improve the local control rate of tumor, control the acute injury of normal tissue and the yield acceptable late treatment-related complications. The specific protocol was as follows: high-risk CTV area (CTV1), 45Gy in total, fraction dose of 1.5Gy, twice a day, bioequivalent dose (BED) of 51.75Gy; Low-risk CTV area(CTV2), 39Gy in total , fraction dose of 1.3Gy, twice a day, BED of 44.07Gy; A total of 30 radiotherapy fraction were performed 10 times a week for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated, histologically confirmed oral cavity carcinoma, staging T2-4N0M0 or T1-4N1-3M0, II-IVB, according to the eighth edition of the AJCC staging system.
2. Pathological evaluation of surgical specimens was pCR (pathologic complete response, no viable tumor cells) or MPR (Major pathologic response, residual viable tumor cells≤10%).
3. Negative surgical margin.
4. No extranodal extension.
5. Aged ≥ 18 years and ≤ 80 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Life expectancy of more than 6 months.
8. Women of childbearing age should agree to the use of contraception (e.g., intrauterine devices, birth control pills, or condoms) during treatment and for 3 months thereafter.
9. The regimen of neoadjuvant therapy can be determined by the clinician.
10. Subjects voluntarily join the study and sign an informed consent form, with good compliance.

Exclusion Criteria:

1. Pregnant or lactating women.
2. A history of other malignant tumors within the previous 5 years or at the time of enrollment, except for cured skin basal cell carcinoma and cervical in situ cancer, as well as thyroid papilloma.
3. Neoadjuvant therapy or radical surgery was not completed.
4. Recurrence or distant metastasis occurred before postoperative radiotherapy.
5. There are contraindications for radiotherapy, chemotherapy, immunotherapy and targeted therapy.
6. Uncontrolled cardiac clinical symptoms or diseases.
7. Serious infections.
8. A history of immunodeficiency, including HIV-positive status or other acquired congenital immunodeficiency diseases, or a history of organ transplantation and bone marrow transplantation.
9. Patients with active tuberculosis infection found by history or CT examination, or patients with active tuberculosis infection history within 1 year prior to enrollment, or patients with active tuberculosis infection history before 1 year without formal treatment.
10. Active hepatitis B (HBV DNA ≥ 2,000 IU/mL or 10,000 copies/mL) or hepatitis C (positive HCV antibody test and HCV RNA above the lower limit of detection).
11. Known history of psychotropic drug abuse, alcoholism and drug use.
12. Not suitable for inclusion, as judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year PFS | 2 years
  PFS is the time from the initiation of therapy to recurrence or death of any cause.

SECONDARY OUTCOMES:
2-year OS | 2 years
  OS is defined as the time interval from the beginning of treatment to death.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial hospital, Sun Yat-sen University, Guangzhou, China